CLINICAL TRIAL: NCT06607172
Title: Antiplaque and Antigingivitis Efficacy of the Combined Effect of Oral Irrigator and Chemicals (0.075% CPC): a Randomized Clinical Trial with Experimental Gingivitis Model
Brief Title: Clinical Efficacy of the Combined Effect of Oral Irrigator and Chemicals (0.075% CPC)
Acronym: WFPOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Federal University of Pelotas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRO 2024-06-WF-POC-BZ-CB
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-09

CONDITIONS: Dental Plaque; Dental Plaque Induced Gingivitis; Dental Plaque and Gingivitis; Gingivitis
Keywords: dental hygiene products; gingivitis; dental plaque; oral irrigator
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Cetylpyridinium

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, examiner blind, parallel-group clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group II: waterflosser + dilutable 0.075% CPC (Active Comparator): Subjects assigned to this group will use a water flosser device and dilutable chemistry product (0.075% CPC) after dilution each time. Water flosser must be used for one minute. They must use this regimen treatment twice daily (in the morning and evening). No other oral hygiene will be allowed during the 21 days of follow-up.
  Interventions: Device: oral irrigator; Drug: Cetylpyridinium Chloride (CPC)
- Group III: negative control (No Intervention): Subjects assigned to this group will abstain for any oral hygiene during the 21 days of follow-up.
- Group I: water flosser and water (Experimental): Subjects assigned to this group will use a water flosser device and water each time. Water flosser must be used for one minute. They must use this regimen treatment twice daily (in the morning and evening). No other oral hygiene will be allowed during the 21 days of follow-up.
  Interventions: Device: oral irrigator

INTERVENTIONS:
Device: oral irrigator — water flosser device
  Arms: Group I: water flosser and water
Device: oral irrigator — water flosser and 0.075% CPC
  Arms: Group II: waterflosser + dilutable 0.075% CPC
Drug: Cetylpyridinium Chloride (CPC) — Cetylpyridinium 0.075%
  Arms: Group II: waterflosser + dilutable 0.075% CPC

SUMMARY:
This is an experimental gingivitis clinical study to evaluate gum health efficacy from the combination effect of water flosser and chemistry (0.075% CPC) compared to water flosser and water and to no oral hygiene regimen with a 3-week follow-up. Thirty participants, aged between 18 and 70, will be enrolled.

DETAILED DESCRIPTION:
This is an examiner blind, randomized controlled, parallel designed clinical study that aims to assess the gum health efficacy (antiplaque and antigingivitis) from the combination effect of water flosser and chemistry (0.075% CPC) compared to water flosser and water and to no oral hygiene in a 3-week experimental gingivitis. Thirty participants will be enrolled and allocated into 3 groups: group I - using a water flosser device and water each time; group II - using a water flosser device and dilutable chemistry product (0.075% CPC) after dilution each time (for groups I an II participants will use this regimen treatment twice daily, in the morning and evening, and no other oral hygiene will be allowed during the 21 days of follow-up); group III - negative control in which participants will abstain for any oral hygiene during the 21 days of follow-up. Gingival index measurements will be the primary efficacy variable after using the assigned regimen for 3 weeks for each subject. Subjects will under go baseline, 3 days, 1, 2 and 3 weeks visits. An Analysis of Covariance will be performed on the final or delta plaque scores using the baseline value as covariate. The F-test in this analysis will test the hypothesis that the waterflosser groups are equal in adjusted means.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Aged between 18 and 70;
* Available for the three (3) week study duration;
* Good general health for participation in the study, based on the opinion of the study investigator;
* Must have at least 20 natural permanent teeth;
* Teeth must meet the scoring entry criteria for dental plaque and gingivitis (gum inflammation) at the discretion of the study examiner.

Exclusion Criteria:

* Medical condition which requires premedication prior to dental visits/procedures;
* Presence of fix/ removable prosthodontics dentures that may interfere with this study clinical examinations;
* Advanced periodontal disease (gum disease) and/or treatment for periodontal disease (including surgery) within the past twelve months;
* Five (5) or more decayed, untreated dental sites (cavities) and/or any dental condition requiring urgent dental care;
* Abnormalities/diseases of the soft or hard oral tissues;
* Orthodontic appliances/bands/lingual bars that interfere with any clinical assessment (plaque scoring)
* Use of drugs that can affect salivary flow;
* Use of antibiotics three (3) months prior to study entry and/or during participation in this study;
* Use of any over the counter medications other than analgesics that could interfere with the study at PI discretion;
* Self-reported pregnancy and/or breastfeeding;
* Current Participation in another clinical study or during the month prior to this clinical study entry;
* Known allergies and/or reactions to common dentifrice ingredients;
* Medical condition which prohibits not eating/drinking or chewing gum for four (4) hours prior to your scheduled visits;
* Immunocompromised conditions (AIDS, immunosuppressive drug therapy);
* Infectious disease and/or other blood borne diseases (Hepatitis series, HIV, tuberculosis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingival Index | 3 weeks
  A Löe-Silness Gingival Index score from 0 to 3 (0 = absence of inflammation and 3 = severe inflammation) will be assigned by the examining dentist to all scorable surfaces of the maxillary and mandibular teeth (6 sites/tooth) using a dental light and dental mirror. A whole mouth mean score for each subject will be determined by adding the values given by the examining dentist to each scorable surface and dividing that number by the total number of surfaces scored.

SECONDARY OUTCOMES:
Navy Plaque Index, Rustogi Modification | 3 weeks
  The dentition will be disclosed with disclosing solution and plaque scored according to the Refined Navy Plaque Index. This index includes nine surfaces (marked A-I) examined for plaque after staining. Surfaces A, B, C denote the gingival margin surfaces, surfaces D and F the proximal surfaces. The total plaque score range is 0-9, the range for the gingival margin area is 0-3 and for the proximal area 0-2.

CONTACTS AND LOCATIONS:
Overall Officials: Wilker Muniz, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No